CLINICAL TRIAL: NCT07105306
Title: A Complementary Approach to Asthma Treatment: Buteyko Breathing Technique
Brief Title: Asthma Treatment: Buteyko Breathing Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seçil Beyece İncazli (Other)
Responsible Party: Sponsor-Investigator, Seçil Beyece İncazli, Lecturer (PhD), Vocational School of Health Services, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EGE-ASHYM-SBİ-01
Record Dates: First submitted 2025-07-17; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Asthma
Keywords: Asthma; Buteyko; complementary therap
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buteyko Breathing Training Group (Experimental): Participants in this group will receive a structured training program on the Buteyko breathing technique, consisting of weekly sessions over 6 months. The intervention aims to improve respiratory function and reduce asthma symptoms through controlled breathing exercises.
  Interventions: Other: Buteyko Breathing Technique Training
- Control Group (No Intervention): Standard Care

INTERVENTIONS:
Other: Buteyko Breathing Technique Training — Buteyko Breathing Technique (BBT), developed in the 1950s, which focuses on reducing dysfunctional hyperventilation patterns through breath control and extended breath-holding phases called control pauses
  Arms: Buteyko Breathing Training Group

SUMMARY:
This study aimed to evaluate the effects of BBT training on asthma control, quality of life, and pulmonary function among asthma patients.The findings suggest that BBT may be a potentially effective complementary approach. However, given the small sample size and short follow-up duration, larger studies with longer-term follow-up are necessary to confirm and generalize these results.

DETAILED DESCRIPTION:
According to certain perspectives, hyperventilation plays a significant role in the manifestation of asthma symptoms. The Buteyko Breathing Technique (BBT), which targets dysfunctional breathing patterns, has been reported to reduce symptoms of hyperventilation and associated anxiety in asthmatic individuals.

This study aimed to evaluate the effects of BBT training on asthma control, quality of life, and pulmonary function among asthma patients.

Between June 2018 and June 2019, this randomized controlled trial was conducted at the asthma outpatient clinic of a university hospital. Approximately 450 asthma patients presented during the study period; 36 eligible participants were assessed, 12 were excluded, and the remaining 24 individuals were randomized (block randomization, block size = 4) into an intervention group (n=12) and a control group (n=12). The intervention group received BBT training and daily practice sessions, while the control group received standard breathing education-based on the "Life with Asthma" booklet-including abdominal and diaphragmatic breathing techniques. All participants were evaluated at baseline and at week 6 using the Asthma Control Questionnaire (ACQ), Asthma Quality of Life Questionnaire (AQLQ), and pulmonary function tests (FEV₁, FEV₁/FVC, control pause (CP)). Data were analyzed using SPSS 25.0; independent t-tests, Mann-Whitney U tests, and repeated-measures ANOVA were applied.

ELIGIBILITY:
Inclusion criteria included patients who:

* were followed in the asthma outpatient clinic of the university hospital,
* had stable asthma (no exacerbation in the last 6 weeks),
* had no communication problems,
* had no history of smoking,
* were using inhaled corticosteroids regularly (without dose changes in the past 4 weeks),
* voluntarily agreed to participate in the study.

Exclusion criteria were as follows:

* presence of another chronic pulmonary disease (e.g., COPD, bronchiectasis),
* psychiatric illness history or use of psychiatric medications,
* cognitive impairment or inability to follow instructions,
* pregnancy or breastfeeding,
* participation in another clinical trial simultaneously.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Change in Asthma Control | Baseline to 6 months after intervention
  Asthma control will be assessed using the Asthma Control Questionnaire (ACQ-6). Higher scores indicate worse control. Scores range from 5 to 25, with lower scores indicating better asthma control. The original Cronbach's alpha was reported as 0.85; in this study, the internal consistency was calculated as 0.88.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared due to ethical and privacy concerns.